CLINICAL TRIAL: NCT06868147
Title: Long-term Clinical and Radiographic Results of Revision Anterior Cruciate Ligament Reconstruction Using Over The Top Single-bundle Technique and Lateral Extra-articular Tenodesis With Achilles Tendon Allograft.
Brief Title: Long-term Clinical and Radiographic Results of Revision Anterior Cruciate Ligament Reconstruction Using a Single-bundle Technique and External Tenodesis With Achilles Tendon Allograft.
Acronym: ACL_REVISION
Status: Recruiting | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Other Study IDs: ACL_REVISION_SBLP
Record Dates: First submitted 2025-03-05; First posted 2025-03-10 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: ACL; LET

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Several techniques for revision of anterior cruciate ligament (ACL) reconstruction and different types of grafts have been used over the years. These include single-bundle techniques, double-bundle techniques, and single-bundle techniques with external tenodesis. We also distinguish between the use of autografts and grafts from donors, or allografts.

The choice of surgical technique and graft type is strongly influenced by the progression of damage characterizing these patients (meniscal, chondral, or ligamentous), the surgical decisions made during the initial surgery (graft used, orientation, and number of bone tunnels), or any complications that occurred.

The use of a specific type of graft is heavily dependent on its availability: it is likely that the first-choice graft for some surgeons may be unavailable because it has already been used. The use of allografts is now commonly accepted by the scientific community, with the Achilles tendon standing out for its biomechanical properties and size. Unlike autografts, it does not damage the patient's ligamentous tissue, which is thus preserved.

Since osteoarthritis is one of the most debated consequences of anterior cruciate ligament revision, an analysis of the results is essential to provide a clearer understanding of the risks and benefits associated with the different types of procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 50 years at the time of surgery;
2. Male and female gender;
3. Patients who have undergone revision of anterior cruciate ligament reconstruction with a single-bundle "Over-The-Top" technique and external tenodesis using Achilles tendon allograft, with or without associated procedures, at least 2 years post-surgery;
4. A radiograph taken immediately before or after the surgery of the affected knee;
5. Patients who have provided consent to participate in the study.

Exclusion Criteria:

1. Patients no longer accessible;
2. Patients who deny consent to participate in the study;
3. Advanced knee osteoarthritis (Outerbridge grade III-IV) at the time of surgery;
4. Severe obesity (BMI > 35);
5. Lower limb conditions that prevent the patient from maintaining an upright position with full weight-bearing during the assessment;
6. Infection or hematological or rheumatic conditions at the time of the assessment.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients will be recruited from all subjects who underwent revision of anterior cruciate ligament reconstruction with the single-bundle "Over-The-Top" technique and external tenodesis using Achilles tendon allograft at the SC Orthopedic and Traumatology Clinic II of the Rizzoli Orthopedic Institute, at least 2 years after the surgical procedure and the clinical-radiological reassessment proposed in this study, between 1/1/2000 and 31/12/2022 at the Rizzoli Orthopedic Institute. This reassessment is part of standard clinical practice.
Sampling Method: Probability Sample
Enrollment: 59 (Estimated)
Dates: Start 2025-03-19 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Lysholm Knee Score | At least 24 months after surgery
  It is a validated measurement scale that assesses knee functionality through 8 items, allowing the evaluation of the knee's condition in relation to the functional demands of daily activities. This assessment tool is used to evaluate the outcomes of surgery in patients who have undergone surgery for ligamentous or meniscal knee injuries. The final score is obtained by summing the various scores from the different items, ranging from 0 to 100. The scores are divided into subgroups: Excellent (95-100); Good (84-94); Fair (65-83); Poor (<64).

SECONDARY OUTCOMES:
Physical examination | At least 24 months after surgery
  A standard physical examination will be performed, and the classic painful points related to meniscal pathology will be assessed.
Anterior drawer test | 24 months after surgery
  it allows the assessment of the anterior translation of the tibia relative to the femur with the knee flexed at 90 degrees. An increase in this translation suggests a lesion of the neo-ACL. It is quantified on a scale from 0 to 3.
Lachman test | At least 24 months after surgery
  it allows the assessment of the anterior translation of the tibia relative to the femur with the knee flexed at 30 degrees. An increase in this translation suggests a lesion of the neo-ACL. It is quantified on a scale from 0 to 3.
Pivot shift test | At least 24 months after surgery
  it is a clinical maneuver used to assess the rotational instability of the knee under examination. The test is performed by applying a stress in internal rotation-valgus and flexion; the occurrence of a "shift" or "clunk" of the tibia suggests a lesion of the neo-ACL associated with rotational instability. It is quantified on a scale from 0 to 3.
International Knee Documentation Committee (IKDC) | At least 24 months after surgery
  The IKDC form is a subjective knee assessment tool that expresses the limitations in the activities the individual can perform in daily life and sports, as well as the presence or absence of symptoms. The three main domains of the IKDC assessment form are: Symptoms, which include pain, stiffness, swelling, and a feeling of locking; Sports and daily activities; Current knee function and function before the injury.
VAS | At least 24 months after surgery
  It is a 10-point unidimensional quantitative pain assessment scale; the scale requires the patient to select the number that best describes the intensity of their pain, from 0 to 10, at that specific moment. 0 means no pain, and 10 indicates the worst possible pain.
Tegner score | At least 24 months after surgery
  It allows the estimation of a subject's level of physical activity with a score between 0 and 10, where 0 represents 'incapacity' and 10 represents 'participation in competitive sports, such as national or international-level football.' This score is the most commonly used to define the level of physical activity in patients with knee disorders. In the study, the Tegner Score will be completed directly by the investigator through an interview with the patient.
PASS score | At least 24 months after surgery
  In order to assess the patient's level of satisfaction, they will be asked to answer the question "Are you satisfied with the surgical intervention?" The response will be dichotomous.
Weight-bearing X-ray of the operated knee (Kellgren-Lawrence scale). | At least 24 months after surgery
  For the radiographic assessment, the patient's clinical and radiological data will be collected, and if necessary, X-rays will be performed to evaluate the development and degree of osteoarthritis, using the Kellgren-Lawrence scale. This scale classifies osteoarthritis into 5 grades, from no arthritic changes (grade 0) to severe joint space narrowing and osteophyte formation (grade 4).
KT-1000 | At least 24 months after surgery
  The KT-1000 is an objective assessment tool that measures the anterior tibial translation relative to the femur's position by applying a predefined force to push the tibia forward. It is commonly used in research to quantitatively assess the static laxity of the knee in the anteroposterior direction after anterior cruciate ligament reconstruction surgeries.
KYRA | At least 24 months after surgery
  KYRA is a non-invasive, outpatient device that allows the assessment of dynamic laxity during the pivot shift phenomenon. The device quantifies the degree of laxity with extreme precision. The unit of measurement is millimeters per square second.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Istituto Ortopedico Rizzoli, Bologna, Italy